CLINICAL TRIAL: NCT05239416
Title: Fat Grafting in Reducing Recurrence in Patients With Healed Venous Ulcers: A Prospective Randomised Clinical Pilot Study
Brief Title: Fat Grafting in Reducing Recurrence in Patients With Healed Venous Ulcers A Prospective Randomised Clinical Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Ireland, Galway, Ireland (Other)
Responsible Party: Principal Investigator, Mohamed Elsharkawi, Mr, National University of Ireland, Galway, Ireland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 118/12
Record Dates: First submitted 2022-01-24; First posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Varicose Ulcer
Keywords: venous, ulcers, fat graft, adipose, stem cells
MeSH Terms: conditions — Varicose Ulcer; Ulcer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fat grafting combined with compression therapy (Experimental): Fat grafting + compression bandages/stockings
  Fat grafting:
  For the purposes of this study, the standard technique will be used for all patients
  * General or local anaesthesia.
  * Performed under the supervision of a plastic surgeon.
  * Harvest site will be either abdomen or lower limb.
  * After harvesting fat by liposuction, the lipoaspirate (which contains the ASCs) will be injected at the base of the healed venous ulcer within the same aseptic operative setting.
  Compression therapy:
  compression bandages / stockings as per routine practice
  Interventions: Procedure: Fat grafting
- Compression therapy only (No Intervention): Compression therapy:
  compression bandages / stockings as per routine practice

INTERVENTIONS:
Procedure: Fat grafting — Under general or local anaesthesia, fat will be harvested from either abdomen or lower limb. After harvesting the fat by liposuction, the lipoaspirate will be injected underneath the healed ulcer area under complete aseptic operative setting
  Arms: Fat grafting combined with compression therapy

SUMMARY:
In this study, investigators aim to use fat grafting in patients with previously healed venous ulcers to study its role on increasing skin thickness and reconstructing skin layers which was damaged by venous hypertension and determine its impact on reducing recurrence rates at 1 year

DETAILED DESCRIPTION:
Study design:

This is a randomised, prospective, active-control pilot study to compare the effectiveness of fat grafting combined with compression therapy to compression therapy alone on reducing ulcer recurrence in patients with healed venous ulcers in a tertiary vascular care centre. This study will randomise 20 patients with previously healed venous ulcers in an equal ratio to one of two treatment arms. The intervention arm will be randomised to undergo fat grafting combined with compression therapy. The control arm will be offered compression therapy only. They will then be followed up in the outpatient clinic at 4 weeks, 8 weeks and 1 year.

Study setting:

Potential participants will be identified and screened at the vascular outpatient clinics within the Saolta group university hospitals, Ireland. Patients will receive the intervention in operating theatre in Roscommon University Hospital (RUH). Fat grafting will be performed under the supervision of a plastic surgeon. The coordinating centre will be the Department of Vascular and Endovascular Surgery, University College Hospital Galway (UCHG), and the School of Medicine at the National University of Ireland Galway (NUI Galway).

Study screening:

Patients with healed venous ulcers will be invited to join the study. Researchers will screen the patient for inclusion and exclusion criteria. Invited patients will be provided with a pre-designed information leaflet. This leaflet will be fully explained to the patient at the initial assessment. The study researchers will answer any questions about the study. Informed consent will be obtained from the patient on a formatted consent form. Patients will be given the freedom to give consent either on the same day or later.

Baseline visit:

Patients will undergo detailed clinical assessment by the researcher as part of the baseline evaluation. Recorded assessments will include:

* Demographics
* General clinical details (ABPI, comorbidities, medication history)
* Previous ulcer history (location, size, time since healing).
* Details of venous disease (previous deep vein thrombosis, previous venous interventions, CEAP classification)
* Assessment and recording skin thickness of the previously healed ulcer area using ultrasound.
* Quality of life and pain scale assessment scores

Sample size:

There are currently no previous studies from which we can withdraw a power calculation for this trial. Previous studies on the use of fat grafting have looked at fat grafting in pressure sores not venous ulcers. To our knowledge there are no studies that have used fat grafting in healed venous ulcers. As such this study is designed as a pilot study. The proposed sample size for this pilot study is 20 patients, being randomised to 10 patients in each arm.

Randomisation:

After meeting the inclusion criteria, screened patients will be randomised to one of two treatment arms. The intervention arm will receive fat grafting combined with compression therapy. The control arm will be offered compression therapy only. This is an intention to treat designed study, where patients are analysed as randomised. Each screened patient will be given a unique screening number.

Sequence generation:

Screened patients will be randomised in a 1:1 ratio of study intervention: control according to a randomisation scheme. The randomisation scheme will be produced using the PROC PLAN® procedure of the SAS® software package (version 9.2.2) using a simple randomisation strategy. The scheme will be concealed from all patients and study personnel until after database lock.

Allocation concealment:

Patients will be allocated to intervention via sequentially numbered opaque sealed envelopes, which will not deliver the randomised allocation except after registering the subject screening number. Each screened patient who is recruited to the trial will be given a unique patient trial number.

Blinding:

It will be impossible to blind the investigator and the patient due to the obvious difference in the surgical approach. Outcome assessors will be blinded. However, in the event of an adverse event outcome assessors will be unblinded.

Statistical analysis:

All data will be analysed according to the intention to treat principle. The comparison of the time to recurrence in the two arms will be performed by using Kaplan Meier survival curves and Log rank test. The outcome measures of recurrence rates and adverse events will be assessed using Chi square or Fisher's Exact, where appropriate. An exact 95% confidence interval will be applied for the difference between intervention groups. Skin thickness will be reported as change from baseline in millimetres. Recurrence rates will be correlated to change in skin thickness

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or more.
* Able to provide written informed consent.
* Healed primary venous ulcers (C5 on CEAP classification) of 5cm or less for at least 1 month.
* Ankle-brachial pressure index (ABPI) of 0.8 or more.

Exclusion Criteria:

* Healed recurrent venous ulcers
* Evidence of deep venous occlusion
* Malignancy or immune-suppression
* Malnutrition
* Multi-organ failure
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Patient's quality of life post fat grafting | 1 year
  Chronic Lower Limb Venous Insufficiency Questionnaire - 14 (CIVIQ-14)

SECONDARY OUTCOMES:
Skin thickness changes | 1 year
  Measured by ultrasound
Recurrence rates | 1 year
  Defined as proportion of new onset break down of epithelium in a fully healed index ulcer within 12 months post intervention
Time to recurrence | 1 year
  Time spent with freedom from recurrent ulceration
Incidence of adverse events | 1 year
  fat embolism, infection, pain and fat necrosis
Pain severity scores | 1 year
  pain numeric scale (1-10)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Elsharkawi, Principal Investigator — University College Hospital Galway
Locations (1):
- Mohamed Elsharkawi, Galway, Ireland

IPD SHARING:
Plan to Share IPD: No